CLINICAL TRIAL: NCT07172438
Title: A Randomized Controlled Trial to Determine the Effect of Flavor Availability on Abstinence With an Electronic Nicotine Delivery System in Primary Combustible Cigarette Smokers.
Brief Title: A RCT to Determine the Effect of ENDS Flavor Availability on Abstinence Within Smokers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RAI Services Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PHCB3US20256
Record Dates: First submitted 2025-09-05; First posted 2025-09-15 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2025-10

CONDITIONS: Smoking; Tobacco
Keywords: Tobacco Harm Reduction; Smoking; Tobacco Use; Tobacco Smoking
MeSH Terms: conditions — Smoking; Tobacco Use; Tobacco Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Tobacco, Menthol, Non Tobacco Non Menthol Flavors (Active Comparator): Participants can choose between tobacco, menthol, and non-tobacco non-menthol flavor variants at one nicotine level (5%).
  Interventions: Other: P2611222; Other: P2615022; Other: P2615122; Other: P2613422
- Tobacco and Menthol Flavor (Active Comparator): Participants can choose between tobacco and menthol flavor variants at one nicotine level (5%).
  Interventions: Other: P2611222; Other: P2613422
- Tobacco Flavor (Active Comparator): Participants can use a tobacco flavor variant at one nicotine level (5%).
  Interventions: Other: P2613422

INTERVENTIONS:
Other: P2611222 — Menthol flavor
  Arms: Tobacco and Menthol Flavor; Tobacco, Menthol, Non Tobacco Non Menthol Flavors
Other: P2615022 — Non-tobacco non-menthol flavor
  Arms: Tobacco, Menthol, Non Tobacco Non Menthol Flavors
Other: P2615122 — Non-tobacco non-menthol flavor
  Arms: Tobacco, Menthol, Non Tobacco Non Menthol Flavors
Other: P2613422 — Tobacco flavor

SUMMARY:
The overall purpose of this study will be to assess primary combustible cigarette users' abstinence from smoking their usual brand of combustible cigarettes at the end of the study, when provided with an electronic nicotine delivery system (ENDS) power unit (2) and varying levels of access to tobacco-flavored, menthol-flavored, or non-tobacco/non-menthol-flavored cartridge-based e-liquids (collectively referred to as the investigational product) within their assigned study arm over a three-month (ninety-day) period.

DETAILED DESCRIPTION:
This will be a multi-site, open-label, randomized controlled trial to evaluate the rate of end-of-study abstinence of healthy adult consumers of combustible cigarettes when provided an electronic nicotine delivery system over a three-month (ninety-day) ambulatory study period.

Potential participants will be recruited and enrolled at 27 sites across the United States. Ipsos will recruit participants in person (e.g., through mall intercepts) at each site or by telephone from existing databases of previous research participants. Based on meeting eligibility requirements, participants will be required to read and sign an Informed Consent Form and to attend a site visit to complete enrollment.

At the Enrollment Visit, participants will be randomized to one of the three study arms. All participants will begin the study with a one-week Trial Period. This Trial Period will allow participants to sample the available flavor(s) within their assigned study arm.

All participants will attend mandatory follow-up site visits on Day 0, Day 30, Day 60, and Day 90, with the option of changing to a different flavor among the available flavors based upon their assigned study arm, if applicable. In the first four weeks of the study, participants in Study Arms 1 and 2 may also attend optional site visits on Day 7, Day 14, and Day 21, with the option of changing flavors among those available in their assigned study arm. All site visits will record the number of study investigational product cartridges dispensed, in addition to all used and unused investigational product cartridges returned.

During the three-month ambulatory study period, participants will be free to use the study investigational product and any other tobacco or nicotine products as desired. The electronic nicotine delivery system (Version 2) power unit technology will measure their puffing topography during use (including puff duration and the time interval between puffs). The puffing topography data will be automatically transferred to a secure online database via a Bluetooth transfer application using the provided smartphone.

Participants will be invited to complete daily, weekly, and monthly surveys, using a mobile application installed on the provided smartphone. Surveys will collect data on:

1. The number of cigarettes smoked the previous day
2. Current flavor use
3. Product liking
4. Number of cigarette quit attempts
5. Use of other tobacco or nicotine products
6. Intent to substitute their usual brand combustible cigarettes for the study investigational product (e.g., gradual, complete, or future intent)
7. Social and environmental factors influencing switching intent

At the conclusion of the ambulatory study period, all participants will return to the study sites for a close-out period and will then be discharged from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand, and are willing to sign an Informed Consent Form (ICF) and complete questionnaires written in English
2. Generally healthy male or female, between 21 and 65 years of age, inclusive, at the time of consent
3. All female (assigned at birth) candidate participants who agree during the pre-screener to receive and take a home pregnancy test prior to the SEV, and who affirm at the SEV that they are not pregnant or intending to become pregnant.

   NOTE: Participants who identify as "intersex" or "unknown" during screening, will be offered the opportunity to receive a pregnancy test if they wish to take one.
4. Currently smoke at least 10 cigarettes on smoking days in the past 30 days
5. Smoke cigarettes regularly for at least 12 months
6. Smoke cigarettes on 15 or more of the past 30 days
7. Smoked at least 100 cigarettes in their lifetime prior to the screening and enrollment visit.
8. Must indicate smoking factory-made filtered menthol and/or non-menthol cigarettes as their primary nicotine product (Occasional use of other tobacco- or nicotine-containing products is acceptable)
9. Indicate a willingness to use ENDS
10. Agree to participate in the study and to abide by the study restrictions and requirements, as described in the informed concent form (ICF)

Exclusion Criteria:

1. Female participants who are pregnant or breastfeeding or planning to become pregnant or start breastfeeding within the next 6 months based on self-report.
2. Female participants who self-report not using adequate methods to prevent pregnancy
3. Persons with pacemakers or other embedded electronic medical devices fitted
4. Persons who self-report heart disease, high blood pressure, diabetes, cancer, Chronic Obstructive Pulmonary Disease, emphysema, asthma or other lung/breathing conditions, a previous history of heart attack or stroke, or are taking medication for depression.
5. Persons who self-report they are allergic/sensitive to cosmetics or fragrances or to any ingredient listed in Vuse commercial products or similar products, including those listed below:

   1. Carvone (L-)
   2. Benzyl alcohol
6. Participants who have used ENDS, nicotine pouch or smokeless tobacco (i.e., chewing tobacco, snus, or snuff) products on 5 or more days in the past 30 days
7. Participants who have used ENDS, nicotine pouch or smokeless tobacco products more than 100 times in their lifetime
8. Participants who have used a nicotine replacement therapy (NRT) product or a prescription drug to help stop smoking (e.g., varenicline, bupropion) in the past 30 days.
9. Employee of a company that manufactures tobacco or ENDS products
10. Persons who are personally, have household members, or have close family or friends in litigation with a company that manufactures tobacco or ENDS products
11. Have taken part in a tobacco/nicotine research study in the past 30 days

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1950 (Estimated)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Past 7-day abstinence from combustible cigarette smoking for the final 7 days of the 13-week study period | 13-weeks
  The odds (i.e., relative probabilities) of participants self-reporting 7-day point prevalence abstinence from combustible cigarette (CC) smoking, as recorded in an electronic diary (eDiary) during the final 7 days of the 13-week study period, comparing Study Arm 1 versus Study Arm 3, and Study Arm 2 versus Study Arm 3.

SECONDARY OUTCOMES:
Odds of final 7-day abstinence between each of the preferred flavor groups (Study Arms 1 and 2). | 13-weeks
  Odds of self-reported final 7-day point prevalence abstinence from combustible cigarette smoking between preferred flavor groups (Study Arms 1 and 2), assessed via electronic diary (eDiary)
Odds rate of final 7-day complete switching between each of the preferred flavor groups (Study Arms 1 and 2 only). | 13-weeks
Time to first 7-day abstinence by Study Arm. | 13-weeks
Time to first 7-day abstinence by preferred flavor group. | 13-weeks
Weekly mean percent cigarettes per day reductions from baseline by Study Arm and preferred flavor group. | 13-weeks
Odds of 50% average weekly cigarettes per day reduction from baseline to final 7-days of study between Study Arm 1 and Study Arm 3, and between Study Arm 2 and Study Arm 3. | 13-weeks
  Odds of achieving ≥50% reduction in average self-reported cigarettes per day (CPD) from baseline to final 7 days of the study, based on daily entries in an electronic diary (eDiary), comparing Study Arm 1 vs. Arm 3 and Arm 2 vs. Arm 3

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Tapia, Ph.D., Study Director — RAIS Service Co
Locations (26):
- United States (26):
  - CRG Test America-Phoenix, Chandler, Arizona
  - C&C-Fort Smith, Fort Smith, Arkansas
  - Research America Orlando, Altamonte Springs, Florida
  - C&C-Tampa, Clearwater, Florida
  - Sago Orlando, Maitland, Florida
  - CRG Test America-Pembroke Pines, Miami, Florida
  - CRG Test America-Ormond Beach, Ormond Beach, Florida
  - C&C-Plantation, Plantation, Florida
  - C&C-Sebring, Sebring, Florida
  - C&C-Tallahassee, Tallahassee, Florida
  - CRG Test America-Tampa, Tampa, Florida
  - C&C-Lombard, Lombard, Illinois
  - C&C-Troy, Troy, Michigan
  - CRG Test America-St. Peters, City of Saint Peters, Missouri
  - C&C-Richmond Heights, St Louis, Missouri
  - Sago St. Louis, St Louis, Missouri
  - Sago Philadelphia, Philadelphia, Pennsylvania
  - C&C-Philadelphia, Philadelphia, Pennsylvania
  - Southern Solutions Knoxville, Knoxville, Tennessee
  - C&C-Arlington, Arlington, Texas
  - Sago Dallas, Dallas, Texas
  - CRG Test America-Grapevine, Grapevine, Texas
  - Sago Houston, Houston, Texas
  - C&C-Humble, Humble, Texas
  - C&C-Mesquite, Mesquite, Texas
  - C&C-San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No